CLINICAL TRIAL: NCT00443560
Title: A Retrospective Case-controlled Study of the Association Between Request to Discontinue Second Stage Labor Epidural Analgesia and Risk of Instrumental Vaginal Delivery
Brief Title: The Association Between Decreasing Labor Analgesia Epidural Infusion and Forceps Delivery
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cynthia Wong, Professor of Anesthesiology, Northwestern University
Other Study IDs: 0524-028
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-03

CONDITIONS: Labor Pain; Pregnancy
Keywords: Labor; Epidural Analgesia; delivery; vacuum extraction; obstetrical Forceps
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Instrumental Vaginal Delivery (IVD): Instrumental vaginal delivery (IVD) is attempted to prevent fetal hypoxia if the second stage of labor is prolonged. It includes forceps and vacuum extractions.
  Interventions: Other: Case controlled analysis of epidural labor analgesia patterns
- Spontaneous Vaginal Delivery (SVD): The control group consisted of parturients who had a spontaneous vaginal delivery (SVD)in the same 24 hour period who were case-matched for gravidity and parity.
  Interventions: Other: Case controlled analysis of epidural labor analgesia patterns

INTERVENTIONS:
Other: Case controlled analysis of epidural labor analgesia patterns — A retrospective study utilizing the Obstetric Anesthesiology Database to identify parturients who received neuraxial labor analgesia initiated with a combined spinal epidural (CSE) technique and maintained with a continuous epidural infusion with patient controlled epidural analgesia boluses
  Other Names: combined spinal epidural analgesia; epidural labor analgesia; bupivacaine; fentanyl

SUMMARY:
The objective of this study will be to compare epidural infusion management, specifically looking at infusion rate changes, in patients who receive forceps deliveries versus normal spontaneous vaginal deliveries. We will match patients based on time and date of delivery, as well as parity, in order to eliminate these variables as potential con-founders.

We hypothesize patients who require a decrease in their basal labor analgesia epidural infusion rate will have an increased incidence of forceps delivery.

DETAILED DESCRIPTION:
The obstetrical anesthesia database will be queried for all forceps deliveries between the dates of January 2004-October 2005. To minimize the influence of different anesthetic and obstetric care providers, the control group consisted of parturients who has spontaneous vaginal deliveries (SVD) in the same 24 hour period who were case-matched for gravidity and parity. Parturients with twin deliveries and fetal demise were not selected for either group.

The database will be queried for the following: maternal age, parity, gestational age, type of analgesia, changes in epidural infusion rate and/or concentration, and supplemental bolus doses of local anesthesia. The data will be stripped of identification by the database manager and entered into a secured computer which is password protected and maintained in the Department of Anesthesiology. The primary endpoint is to evaluate if decreasing the epidural infusion rate was associated with a forceps delivery.

ELIGIBILITY:
Inclusion Criteria:

* Singletons
* Viable fetal vaginal deliveries between January 2004-October 2005

Exclusion Criteria:

* Outside specified time frame
* Multiparity
* Fetal demise

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women
Sampling Method: Probability Sample
Enrollment: 2162 (Actual)
Dates: Start 2006-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Wong, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Murphy DJ. Failure to progress in the second stage of labour. Curr Opin Obstet Gynecol. 2001 Dec;13(6):557-61. doi: 10.1097/00001703-200112000-00002. PMID 11707657
- [Background] Comparative Obstetric Mobile Epidural Trial (COMET) Study Group UK. Effect of low-dose mobile versus traditional epidural techniques on mode of delivery: a randomised controlled trial. Lancet. 2001 Jul 7;358(9275):19-23. doi: 10.1016/S0140-6736(00)05251-X. PMID 11454372
- [Background] Torvaldsen S, Roberts CL, Bell JC, Raynes-Greenow CH. Discontinuation of epidural analgesia late in labour for reducing the adverse delivery outcomes associated with epidural analgesia. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD004457. doi: 10.1002/14651858.CD004457.pub2. PMID 15495111
- [Background] Hess PE, Pratt SD, Soni AK, Sarna MC, Oriol NE. An association between severe labor pain and cesarean delivery. Anesth Analg. 2000 Apr;90(4):881-6. doi: 10.1097/00000539-200004000-00020. PMID 10735793
- [Background] Cohen SE, Yeh JY, Riley ET, Vogel TM. Walking with labor epidural analgesia: the impact of bupivacaine concentration and a lidocaine-epinephrine test dose. Anesthesiology. 2000 Feb;92(2):387-92. doi: 10.1097/00000542-200002000-00019. PMID 10691224
- [Background] Panni MK, Segal S. Local anesthetic requirements are greater in dystocia than in normal labor. Anesthesiology. 2003 Apr;98(4):957-63. doi: 10.1097/00000542-200304000-00024. PMID 12657859
- [Background] Yancey MK, Zhang J, Schweitzer DL, Schwarz J, Klebanoff MA. Epidural analgesia and fetal head malposition at vaginal delivery. Obstet Gynecol. 2001 Apr;97(4):608-12. doi: 10.1016/s0029-7844(00)01230-8. PMID 11275036
- [Background] Wong CA, Scavone BM, Peaceman AM, McCarthy RJ, Sullivan JT, Diaz NT, Yaghmour E, Marcus RJ, Sherwani SS, Sproviero MT, Yilmaz M, Patel R, Robles C, Grouper S. The risk of cesarean delivery with neuraxial analgesia given early versus late in labor. N Engl J Med. 2005 Feb 17;352(7):655-65. doi: 10.1056/NEJMoa042573. PMID 15716559
- [Background] 9. Wong CA, Scavone BM, Sullivan JT, Ebarvia MJ, McCarthy RJ. The risk of cesarean delivery with early neuraxial analgesia in nulliparous induction of labor. http://www.asa-abstracts.com 2007:A1204.
- [Background] Ben-Haroush A, Melamed N, Kaplan B, Yogev Y. Predictors of failed operative vaginal delivery: a single-center experience. Am J Obstet Gynecol. 2007 Sep;197(3):308.e1-5. doi: 10.1016/j.ajog.2007.06.051. PMID 17826432
- [Background] Ziadeh S, Yahaya A. Pregnancy outcome at age 40 and older. Arch Gynecol Obstet. 2001 Mar;265(1):30-3. doi: 10.1007/s004040000122. PMID 11327090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Obstetric Anesthesiology Database was used to identify parturients from the Labor and Delivery Unit of Prentice Women's Hospital of Northwestern Memorial Hospital who qualified for the study between January 2004 and October 2005.
Period: Overall Study
Arm/Group | Instrumental Vaginal Delivery (IVD) | Spontaneous Vaginal Delivery (SVD)
Started | 1081 | 1081
Completed | 1021 | 1051
Not Completed | 60 | 30
Not completed — No intrathecal dose | 58 | 26
Not completed — Multiple pregnancies or fetal demise | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Instrumental Vaginal Delivery (IVD) | Spontaneous Vaginal Delivery (SVD) | Total
Number analyzed (Participants) | 1081 | 1081 | 2162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1081 | 1081 | 2162
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (3) | 31 (3) | 31 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1081 | 1081 | 2162
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1081 | 1081 | 2162

OUTCOME MEASURES:

1. Primary Outcome: Number of Parturients With a Decrease in the Infusion of Epidural Analgesia During Second Stage of Labor
Description: At the request of the obstetric provider, second stage analgesia density was decreased by decreasing the basal infusion rate if there was dissatisfaction with the progress of labor or a perceived inability to push. The basal infusion was never totally discontinued.
Time Frame: Second stage of labor up to 3 hours
Population: Analysis was per protocal
Measure: Number; unit: participants
Arm/Group | Instrumental Vaginal Delivery (IVD) | Spontaneous Vaginal Delivery (SVD)
Number analyzed (Participants) | 1021 | 1051
participants | 146 | 51
Statistical Analysis 1: Comparison: Instrumental Vaginal Delivery (IVD) vs Spontaneous Vaginal Delivery (SVD); Test type: Superiority or Other; p < 0.01, Chi-squared, Corrected; Odds Ratio (OR) = 3.3, 95% CI [2.3 to 4.5]

2. Secondary Outcome: Number of Participants With Breakthrough Pain in the First Stage of Labor
Description: Pain not responding to epidural analgesia in the first stage of labor was treated with bolus dose of bupivacaine 1.25 mg/mL or lidocaine 10 mg/mL, 10 to 15 mL. If pain relief was obtained the infusion concentration was increased. If the patient had no pain relief following the bolus injection, the epidural catheter was replaced.
Time Frame: Supplemental analgesia in first stage of labor (<24 hours)
Population: Analysis was per protocol
Measure: Number; unit: participants
Arm/Group | Instrumental Vaginal Delivery (IVD) | Spontaneous Vaginal Delivery (SVD)
Number analyzed (Participants) | 1021 | 1051
participants
  Supplemental bolus | 802 | 243
  Infusion increase | 149 | 87
  Concentration increase | 32 | 19
Statistical Analysis 1: Comparison: Instrumental Vaginal Delivery (IVD) vs Spontaneous Vaginal Delivery (SVD); Test type: Superiority or Other; p < 0.01, Chi-squared, Corrected; Odds Ratio (OR) = 12.2, 95% CI [9.9 to 15.0]

3. Secondary Outcome: Duration of Labor Analgesia
Description: Time in minutes from initiation of labor analgesia until delivery of the infant
Time Frame: Time form initiation of labor analgesia to delivery (up to 24 hours)
Population: Analysis was per protocal
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Instrumental Vaginal Delivery (IVD) | Spontaneous Vaginal Delivery (SVD)
Number analyzed (Participants) | 1021 | 1051
minutes | 420 [300 to 570] | 300 [210 to 420]
Statistical Analysis 1: Comparison: Instrumental Vaginal Delivery (IVD) vs Spontaneous Vaginal Delivery (SVD); Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Description: Adverse events were not extracted from charts reviewed in this study
Arm/Group | Instrumental Vaginal Delivery (IVD) | Spontaneous Vaginal Delivery (SVD)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The retrospective design incurs the risk of unrecorded or unobserved data. The sample selected included all patients with neuraxial analgesia who underwent IVD, but a limited sample of SVD.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes